CLINICAL TRIAL: NCT04619329
Title: Safety and Efficacy of GSMs-TACE Combined With Surgical Resection in Treatment of Huge Hepatocellular Carcinoma (HCC) (≥10cm): A Single Center, Open, Randomized Controlled Trial.
Brief Title: Safety and Efficacy of GSMs-TACE Combined With Surgical Resection in Treatment of Huge Hepatocellular Carcinoma (HCC) (≥10cm)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200-0-02
Record Dates: First submitted 2020-11-03; First posted 2020-11-06 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Huge Hepatocellular Carcinoma (HCC) (≥10cm)
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSMs-TACE+ Surgical Resection Group (Experimental): After TACE using Lobaplatin and GSMs (150-350μm, 350-560μm, 560-710μm or 710-1000μm), patients will receive surgical resection 15-30 days later, as specified per protocol.
  Interventions: Device: GSMs-TACE; Procedure: Surgical Resection
- Surgical Resection Group (Active Comparator): Patients will receive surgical resection, as specified per protocol.
  Interventions: Procedure: Surgical Resection

INTERVENTIONS:
Device: GSMs-TACE — TACE using Lobaplatin (30-40mg/m2) and gelatin sponge microspheres (150-350μm, 350-560μm, 560-710μm or 710-1000μm)
  Other Names: TACE
  Arms: GSMs-TACE+ Surgical Resection Group
Procedure: Surgical Resection — Surgical Resection of HCC
  Other Names: Hepatectomy

SUMMARY:
A Single center, Open, Randomized Controlled Trial Evaluating the Safety and Efficacy of GSMs-TACE combined with Surgical Resection in Treatment of Huge Hepatocellular Carcinoma (HCC) (≥10cm).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed imaging and pathological diagnosis of HCC, or diagnosed for the first time according to the guidelines for diagnosis and treatment of primary liver cancer in China (2019 edition).
2. Barcelona Clinic Liver Cancer (BCLC) stage A or B.
3. Remnant liver volume and liver function reserve are suitable for surgical resection.
4. Main lesion diameter ≥10cm.
5. Number of HCC lesions ≤5 and all located on one liver lobe.
6. Liver function Child-Pugh class A
7. ECOG Performance Status 0-1
8. Life expectancy ≥ 6 months
9. HCC is diagnosed for the first time.
10. Age 18 to 75 years
11. Able to sign and provide written informed consent.

Exclusion Criteria:

1. Severe active infection >grade 2 (except for Hepatitis B and C infection).
2. Liver function Child-Pugh class C.
3. BCLC stage C.
4. Patients with unresectable HCC.
5. Platelet <60×109/L.
6. Concomitant malignant tumors in other organs.
7. Patient with severe cardiac, lung or kidney disease, or severe diabetes.
8. Pregnant or breast-feeding woman.
9. Patients with severe neuropathy and unable to report therapeutic effects.
10. Patients with severe atherosclerosis.
11. Patients with AIDS.
12. Severe hemorrhage of digestive tract within the 4 weeks prior to enrolment.
13. Severe thrombogenesis or embolic event within the 6 months prior to enrolment.
14. Currently enrolled or going to enroll in any other clinical trials.
15. Subject is not suitable to participate in the study as judged by investigator (poor patient compliance，inability to follow up).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival（DFS） | 6 months
Median Overall Survival (mOS) | 2 years

SECONDARY OUTCOMES:
Incidence of Intrahepatic Metastasis | 6 months
Incidence of Extrahepatic Metastasis | 1 and 2 years
Overall Survival (OS) | 1 and 2 years
Adverse Events | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Beijing, China